CLINICAL TRIAL: NCT00817921
Title: Effect of Prematurity on Renal Function in 5 Years Old Children Comparison of Former Premature Children Treated by Ibuprofen in the Neonatal Period to Controls
Brief Title: Effect of Prematurity on Renal Function in 5 Years Old Children
Acronym: SUIVIREIN
Status: Completed | Type: Observational
Sponsor: Jean Michel Hascoet (Other)
Responsible Party: Sponsor-Investigator, Jean Michel Hascoet, Professor, Maternite Regionale Universitaire
Organization: Maternite Regionale Universitaire (Other)
Other Study IDs: MRU-07-11
Record Dates: First submitted 2009-01-06; First posted 2009-01-07 (Estimated); Last update posted 2014-02-05 (Estimated); Status verified 2014-02

CONDITIONS: Prematurity of Fetus
Keywords: premature renal function; ibuprofen; blood pressure; Renal function

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood and urine samples
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- 1: former premature children treated by ibuprofen
- 2: former premature children not treated by ibuprofen
- 3: former term children (control)

SUMMARY:
Purpose of the study:

1. To evaluate the effect of prematurity on renal function in 5 years old children
2. To compare former premature children treated by ibuprofen in the neonatal period to controls

ELIGIBILITY:
Inclusion Criteria:

* Former premature children included at birth in a trial about ibuprofen and renal function in premature infants (ClinicalTrial.gov identifier:NCT00217191)

Exclusion Criteria:

* lack of parental consent

Ages: 3 Years to 5 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: children from a previous trial followed at 3, 4 and 5 years of age
Sampling Method: Non-Probability Sample
Enrollment: 168 (Actual)
Dates: Start 2008-11; Primary Completion 2012-12 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Creatinine clearance | 5 years of age

SECONDARY OUTCOMES:
Growth | at 3 years of age
Blood Pressure | 5 years of age
Hemodynamic tolerance to mild exercise | 3 years of age
Growth | 4 years of age
Growth | 5 years of age
Hemodynamic tolerance to mild exercise | 4 years of age
Hemodynamic tolerance to mild exercise | 5 years of age

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Michel HASCOET, MD, Principal Investigator — Maternite Regionale Universitaire
Locations (3):
- France (3):
  - CHU, Dijon
  - AP-HM (Néonatologie), Marseille
  - Maternite Regionale Universitaire, Nancy

REFERENCES:
- [Derived] Vieux R, Hascoet JM, Franck P, Guillemin F. Increased albuminuria in 4-year-old preterm-born children with normal height. J Pediatr. 2012 Jun;160(6):923-8.e1. doi: 10.1016/j.jpeds.2011.12.005. Epub 2012 Jan 18. PMID 22261507